CLINICAL TRIAL: NCT02030106
Title: Revealing the Role of the Cervico-vaginal Microbiome in Spontaneous Preterm Birth
Brief Title: Motherhood and Microbiome
Acronym: M&M
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 818914; R01NR014784-01 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-08 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Preterm Birth
Keywords: Cervicovaginal microbiome; Microbiome; Preterm Birth; Cervical Remodeling; Preterm delivery; Microbiota
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Women will self-collect samples of their cervicovaginal fluid using large cotton swabs.
  Subjects who have had a previous preterm birth will also have cervical cells collected in the same manner that cells are collected for a routine pap smear.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prior Preterm Birth Patients: All obstetrical patients eligible for the study that have had a prior preterm birth.
- Term Birth Patients: All obstetrical patients eligible for the study that have not had a prior preterm birth.

SUMMARY:
This is a prospective cohort, enriched with women with a prior term birth, of singleton pregnancies who will be followed for the outcome of preterm birth. The main exposure of interest is the characterization of the cervico-vaginal microbiota. Women will be recruited from a population seeking routine obstetrical care at obstetrical practices at Penn. They will have three research visits during pregnancy to complete questionnaires and collect samples of cervico-vaginal fluid and cervical cells. Outcome data will be collected about the prenatal events and timing of delivery.

DETAILED DESCRIPTION:
Patients will be recruited around the time of their routine obstetrical visits. They will be asked to participate in three visits total. Visit one/enrollment occurs between 16 and 20 weeks of gestation, visit two at 20-24 weeks, and visit three at 24-28 weeks. At each visit, vaginal swabs will be collected. The patient will also be asked to fill out a series of surveys related to stress, anxiety,and depression in pregnancy. Research coordinators will perform chart abstraction after delivery.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women receiving care in University of Pennsylvania Health System

Exclusion Criteria:

* Non-singleton pregnancy (twins, triplets, etc.)
* Known major fetal anomaly
* Known HIV positive status
* History of organ transplant
* Chronic steroid use (greater than 20 mg per day for more than 30 days at the time of first study visit)

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women will be recruited from three locations: Penn ObGyn Associates, Helen O. Dickens Clinic, and Maternal Fetal Medicine at 2000 Courtyard. Potential subjects will be identified from clinical schedules and will be pre-screened in EPIC for eligibility. They may be approached during a clinical visit, or the research team may call them prior to or after a scheduled visit to introduce the study. Women can be enrolled anytime between the confirmation of pregnancy and 20 weeks/0 days gestation. For convenience, research visits can be conducted at the time of a scheduled clinical visit, or at a separate time.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2013-10; Primary Completion 2017-02-03 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Cervicovaginal Microbiota in Women With and Without Preterm Birth | Enrollment through delivery
  Cervicovaginal Microbiota in Women With and Without Preterm Birth

SECONDARY OUTCOMES:
Potential Modifiers of the Cervicovaginal Microbiome | Enrollment through delivery
  Potential modifiers of the cervicovaginal microbiome: behavioral factors, stress, nutrition/obesity, vaginal infections, genetic or host immune differences, race and ethnicity, social behaviors, environmental influences

CONTACTS AND LOCATIONS:
Overall Officials: Michal A Elovitz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States